CLINICAL TRIAL: NCT01617408
Title: TMS Investigations of the Human Visual System
Brief Title: Brain Stimulation and Vision Testing
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120128; 12-M-0128
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-10-28

CONDITIONS: fMRI; Dorsal Pathway; Ventral Pathway
Keywords: Theta Burst Stimulation; Transcranial Magnetic Stimulation (TMS); Visual Cortex; Visual Processing; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Neurologically normal subjects aged 18 to 50 years old

SUMMARY:
Background:

-The brain has two systems for recognizing objects. One system recognizes what an object is, and the other system recognizes where the object is located. However, there is much about how the brain handles and interprets the information from these two systems that is still unclear. Researchers want to study the parts of the brain that are involved in how vision is processed. They will use magnetic resonance imaging (MRI) and transcranial magnetic stimulation (TMS) or transcranial electrical stimulation (tES) on the brain. MRI measures what parts of the brain become more active when tasks are performed. TMS uses magnetic pulses to temporarily change the activity in parts of the brain. tES uses electrical current to temporarily change brain function.

Objectives:

-To better understand how people visually recognize different types of objects.

Eligibility:

-Healthy volunteers between 18 and 50 years of age, who only speak English.

Design:

* This study includes many different experiments on vision. Each experiment may combine visual tasks, MRI scans, and TMS or tES. Participants may be asked to have several different tests. Each test will require a separate visit to the National Institutes of Health.
* Participants will be screened with a physical exam and medical history. They will have a baseline brain scan at the first visit.
* Participants may do visual tasks alone, with MRI only, with TMS or tES only, or with MRI and TMS or tES combined. For the visual tasks, they will look at pictures of objects on a computer screen. Sometimes the images will appear very briefly (less than one-tenth of a second). Sometimes they will appear for up to 5 seconds. These images will be of things like faces, bodies, tools, and scenes. Participants will be asked to respond in different ways to the pictures. They may respond by typing on a computer keyboard or by pressing a button. Participants will have time to practice the tasks before the experiment.
* Participants will remain on the study for up to 3 years.

DETAILED DESCRIPTION:
Objective

An influential model of cortical organization proposes that the primate visual system is divided into two functionally distinct pathways (Ungerleider & Mishkin, 1982). The ventral or what visual pathway, which projects from occipital cortex into the ventral temporal cortex, is principally used for object recognition and identification. The dorsal or where pathway, which projects from occipital cortex into the parietal cortex, is principally used for locating the position of objects in the visual field and for action planning. In the proposed series of experiments we will investigate how neural representations in the ventral and dorsal pathways contribute to a range of cognitive tasks including object and scene recognition, attentional selection and face processing. These experiments will principally use transcranial magnetic stimulation (TMS) or transcranial electrical stimulation (tES) in combination with functional magnetic resonance imaging (fMRI).

TMS and tES provide unique experimental tools for studies of human cognitive function because they can be used to transiently and safely disrupt or enhance the neural processing in a targeted cortical region while subjects perform concurrent behavioral tasks that depend on the operations of that region. Furthermore TMS and tES can be combined with neuroimaging techniques such as fMRI to examine the remote effects of the induced neural disruption in other task-dependent regions distributed across cortex. We plan to use TMS and tES to address unanswered questions concerning the functioning of the distributed neural networks for different categories of object recognition and in the attention network of the human brain.

Study Population

We plan to test 665 neurologically normal subjects aged between 18 and 50 years old. Subjects will also take part in an fMRI experiment prior to any subsequent TMS or tES experiments in order to localize the stimulation sites of interest.

Design

The aim of the proposed series of experiments is to examine the effects of the TMS and tES induced neural disruption or enhancement on behavioral task performance and the neural correlates of the impaired performance as measured with fMRI. Broadly these experiments can be divided into studies that use online and offline TMS or tES. In on-line experiments, TMS or tES will be applied during behavioral tasks. In off-line experiments, theta burst stimulation (TBS) or tES will be delivered before the experimental task and off-line experiments may combine TBS or tES with fMRI.

1. TMS or tES target site localization

   Prior to both online and offline studies subjects will take part in an fMRI experiment designed to localize particular cortical regions of interest (ROIs). The fMRI experiment will require the subject to view either a series of different object categories (e.g. faces, bodies, scenes) or flickering sections of black and white checkerboards in the fMRI scanner. The results of these fMRI experiments will be used to identify regions of cortex that will then be targeted with TMS or tES. We will identify TMS and tES target sites using the stereotaxic Brainsight co-registration software and the scalp location will be marked individually on each subject.
2. Online behavioral TMS experiments

   Online TMS experiments are designed to address the direct effects of the induced neural disruption on the targeted TMS site only. TMS is delivered during every trial to assess the effects on concurrent task performance. Subjects will perform a range of visual behavioral tasks while online TMS is delivered over the cortical region of interest or over control sites (e.g. vertex). Repetitive TMS will be delivered at a frequency of 10Hz for 500ms. In some experiments we will alternatively deliver double-pulse TMS at different latencies after stimulus onset to assess when the targeted region is likely to be involved in task performance.
3. Offline TBS experiments

   Offline thetaburst (TBS) experiments are also designed to assess the effects of the induced disruption in the stimulated region. However, rather than delivering TMS during every experimental trial Thetaburst TMS (TBS) is delivered over the targeted region of interest (ROI) for latencies up to 60 seconds prior to the subject performing any behavioral task. The neural effects of this induced disruption have then been shown to last for up to 30 minutes (Huang et al., 2005). In the offline TBS experiments we propose to deliver 60 seconds of the TBS over the stimulated ROI. In some of the proposed experiment participants will then be placed in an fMRI scanner before and after TBS stimulation. During both fMRI sessions subjects will perform a series of visual discrimination tasks to assess the effects of TBS disruption both on their behavior and on activity in remote cortical areas as measured with BOLD activation.
4. Online & offline tES experiments

Behavioral impact of tES can be recorded both online and offline simultaneously within the same session and using the same protocol. Online tES examines the direct effect of neural stimulation whilst a participant is performing a task (Tyler et al., 2018). Unlike TMS, online tES is possible as the subcutaneous stimulation effects are minor or unperceived, have no auditory impact, and require no experimenter involvement. Once the surface electrodes are in place, the participant is free to act independently. Offline tES examines the time-course of behavioral impact after stimulation. The offline effects of tES last up to 60 minutes after stimulation (Terney et al., 2008; Herpich et al., 2019). We may deliver either direct or alternating current tES for a maximum of 20 minutes, at an intensity under 4mA (Antal et al., 2017; Rossi & Antal, 2020).

Outcome measures

The dependent variables in the online behavioral TMS or tES experiments will be performance accuracy, sensitivity (d ) and reaction time (RT) measures collected during the concurrently performed behavioral tasks. Dependent variables in the offline fMRI-TBS or fMRI-tES experiments will be task performance as well as reduced neuronal activity as measured by decreased BOLD activation in the targeted and remote ROIs.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy

Ages 18-50 years (inclusive)

Able to read and write in English to guarantee understanding of all written and spoken instructions, which are in English

EXCLUSION CRITERIA:

Individuals with conditions that could pose a risk relating to the safety of the MRI procedure, the TMS procedure or the combined TBS and fMRI procedure will be excluded from the protocol such as:

* Those with ferromagnetic metal in the cranial cavity or eye, e.g. aneurysm clip, implanted neural stimulator, cochlear implant, ocular foreign body.
* Those with an abnormality on a structural MRI.
* Those with an implanted cardiac pacemaker or auto-defibrillator
* Those with an insulin pump.
* Those with an irremovable body piercing
* Pregnant women
* Those with a visual impairment that will prevent them from performing the task
* Those without consent capacity will not be enrolled
* Those who do not understand the study instructions
* Those with a history of neurological problems. Neurological problems include, but are not limited to; family history of epilepsy, history of seizures and recurrent migraines.
* Those using medicines that can lower the seizure threshold. These can include but are not limited to; imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines.
* Those with a visual impairment that will prevent them from performing the task
* Those who have a significant psychiatric illness or have a history of psychiatric illness.
* NIMH staff/employees/family members

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Neurologically normal subjects aged between 18 and 50 years old.
Sampling Method: Non-Probability Sample
Enrollment: 665 (Estimated)
Dates: Start 2013-03-04 (Actual)

PRIMARY OUTCOMES:
Online behavioral TMS experiments: performance accuracy, sensitivity (d') and reaction time (RT); Offline fMRI TBS experiments: task performance as well as reduced neuronal activity | Ongoing
  a. Behavioral TMS or tES experiments will measure the speed of a key press to indicate the correct answer and performance accuracy on the task. b. Offline TMS that combine TBS or tES with fMRI will measure changes in BOLD activation in the targeted region as well as in connected cortical areas identified with an independent localizer.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher I Baker, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aguirre GK, D'Esposito M. Topographical disorientation: a synthesis and taxonomy. Brain. 1999 Sep;122 ( Pt 9):1613-28. doi: 10.1093/brain/122.9.1613. PMID 10468502
- [Background] Amemori K, Sawaguchi T. Rule-dependent shifting of sensorimotor representation in the primate prefrontal cortex. Eur J Neurosci. 2006 Apr;23(7):1895-909. doi: 10.1111/j.1460-9568.2006.04702.x. PMID 16623846
- [Background] Barker AT, Jalinous R, Freeston IL. Non-invasive magnetic stimulation of human motor cortex. Lancet. 1985 May 11;1(8437):1106-7. doi: 10.1016/s0140-6736(85)92413-4. No abstract available. PMID 2860322
- [Derived] Groen IIA, Silson EH, Pitcher D, Baker CI. Theta-burst TMS of lateral occipital cortex reduces BOLD responses across category-selective areas in ventral temporal cortex. Neuroimage. 2021 Apr 15;230:117790. doi: 10.1016/j.neuroimage.2021.117790. Epub 2021 Jan 23. PMID 33497776
- [Derived] Pitcher D, Pilkington A, Rauth L, Baker C, Kravitz DJ, Ungerleider LG. The Human Posterior Superior Temporal Sulcus Samples Visual Space Differently From Other Face-Selective Regions. Cereb Cortex. 2020 Mar 21;30(2):778-785. doi: 10.1093/cercor/bhz125. PMID 31264693
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-M-0128.html